CLINICAL TRIAL: NCT06477952
Title: Targeted Treatment of Obstructive Sleep Apnea With Dronabinol: Proof of Concept and Phase II Clinical Trial
Brief Title: DRonabinol Treatment of OSA
Acronym: DROSA
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of Illinois at Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PULM-011-23F
Record Dates: First submitted 2024-06-21; First posted 2024-06-27 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Obstructive Sleep Apnea
Keywords: OSA; sleep apnea; pharmacological treatment; Drug treatment
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes | interventions — Dronabinol

STUDY DESIGN:
Intervention Model Description: 120 Veterans will be screened and enrolled to achieve 45 participants completing the study. All participants will receive oral Dronabinol treatment nightly for two weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Single group (Experimental): Open label Dronabinol treatment for two weeks.
  Interventions: Drug: Dronabinol

INTERVENTIONS:
Drug: Dronabinol — Open label Dronabinol treatment for two weeks.
  Other Names: Marinol

SUMMARY:
This is an open-label trial that tests the effectiveness of Dronabinol in treating obstructive sleep apnea (OSA). All participants will take oral Dronabinol for two weeks. Sleep studies will be conducted before and after treatment to measure OSA severity.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA), is a serious respiratory disorder that involves repetitive cessation of breathing during sleep. It is estimated that 15-20 million people in the United States suffer from OSAS, which has been linked to increased risk for hypertension, heart failure, depression, and diabetes. The current standard of care for OSA, positive airway pressure (PAP), involves a mechanical device with low patient tolerance and adherence. Upper airway surgical approaches are also an option but are invasive and often unsuccessful. Effective drug treatments for OSA remain to be identified.

This study will enroll up to 120 Veterans so that 45 Veterans may complete the two-week open-label Dronabinol treatment trials. The results of the study will be used to develop a prediction model for OSA severity reduction after 2-week Dronabinol treatment vs. pretreatment AHI. Participants clinical (age, sex, body mass index, comorbidity) and pretreatment polysomnographic characteristics (sleep architecture, respiratory disturbance, and endotypes; loop-gain, arousal threshold, upper airway collapsibility and compensation) will be used to develop a prediction model for improvement of OSA with Dronabinol treatment. This prediction model will be used for a randomized clinical trial after the completion of this trial.

ELIGIBILITY:
Inclusion Criteria:

1. Adults 18 to 65 years of age.
2. AHI 15-50 per hour on pre-treatment polysomnography.

Exclusion Criteria:

1. Positive Airway Pressure (PAP) treatment of OSA: use > 4 hours per day for 30% of days within 3 months of enrollment. PAP use will be determined from device download data.
2. Hypoglossal nerve stimulator (HNS) or oral appliance device treatment with use > 4 hours per day for 30% of days within 3 months of enrollment. HNS use will be determined by device download and oral appliance use by self-report.
3. History of upper airway surgery for OSA (except adenotonsillectomy).
4. Central or mixed apneas >25% of respiratory events on diagnostic polysomnography.
5. Arterial oxygen saturation < 75% for > 5% sleep time on pretreatment polysomnography.
6. Body mass index > 45 kg/m2.
7. If post-bariatric surgery, weight must be stable ±5% (per electronic medical records) for at least 6 months before the first dose of the study drug.
8. Active enrollment in a weight loss program.
9. Shiftwork within 3 months of enrollment.
10. High-risk occupation: commercial driver and pilot.
11. Motor vehicle accident or near-miss incident within 1 year of enrollment.
12. Current drug or habitual alcohol use or positive urine drug screen.
13. Comorbid medical and psychiatric disorders:

    1. Primary sleep disorders: e.g., narcolepsy, restless legs syndrome.
    2. Uncontrolled mood disorder or a diagnosis of schizophrenia.
    3. Initiation of new antidepressant or antipsychotic medication within 3 months.
    4. Identified as high-risk for suicide in electronic health records.
    5. Uncontrolled medical disorders (coronary heart disease, arrhythmia, congestive heart failure, chronic obstructive pulmonary disease, chronic hypoxemic or hypercapnic respiratory failure, stroke within 6 months of enrollment, chronic liver or kidney disease, autoimmune disorders).
14. Use of sedative-hypnotic medications within 30 days of enrollment.
15. Complete blood count or liver function test values more than 1.5 times the upper limit of normal.
16. Pregnancy.
17. Allergy to cannabinoids or sesame oil.
18. Average weekly alcohol consumption of more than 10 servings.
19. Participation in other investigational protocols within 30 days of enrollment.

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Apnea hypopnea index (AHI) | 2 weeks
  The change in AHI after two weeks of Dronabinol treatment will be determined from before and after treatment polysomnograms.

SECONDARY OUTCOMES:
T<90 | 2 weeks
  The change in time below 90% oxygen saturation (T<90) after two weeks of Dronabinol treatment will be determined from before and after treatment polysomnograms.

OTHER OUTCOMES:
Psychomotor Vigilance Test (PVT) | 2 weeks
  The change in Lapses on Psychomotor Vigilance Test (PVT) after two weeks of Dronabinol treatment will be determined from before and after treatment PVT using a 10 minute protocol.
24-hour mean arterial blood pressure (BP) | 2 weeks
  The change in 24- hour mean arterial blood pressure after two weeks of Dronabinol treatment will be determined from before and after treatment 24-hiur ambulatory BP recording.
Sleep Efficiency | 2 weeks
  The change in sleep efficiency after two weeks of Dronabinol treatment will be determined from before and after treatment polysomnograms.
REM sleep | 2 weeks
  The change in REM sleep after two weeks of Dronabinol treatment will be determined from before and after treatment polysomnograms.
Slow wave sleep | 2 weeks
  The change in slow wave sleep after two weeks of Dronabinol treatment will be determined from before and after treatment polysomnograms.
Treatment Satisfaction Questionnaire for Medication (TSQM) | 2 weeks
  Patient reported treatment satisfaction. TSQM scores have a range of 0 to 100, with higher scores indicating higher satisfaction.
Epworth Sleepiness Scale (ESS) | 2 weeks
  The change in Epworth Sleepiness Scale (ESS) will be measured after two weeks of Dronabinol treatment.
  ESS scores have a range of 0 to 24, with higher scores indicating greater sleepiness.
Functional Outcomes of Sleep Questionnaire (FOSQ) | 2 weeks
  The change in Functional Outcomes of Sleep Questionnaire (FOSQ) will be measured after two weeks of Dronabinol treatment.
  FOSQ score ranges from 5-20, with higher scores indicating better functional status.
Pittsburgh Sleep Quality Index (PSQI) | 2 weeks
  The change in Pittsburgh Sleep Quality Index (PSQI) will be measured after two weeks of Dronabinol treatment.
  The PSQI score ranges from 0 to 21. Higher scores indicate poorer sleep quality.
Insomnia Severity Index (ISI) | 2 weeks
  The change in Insomnia Severity Index (ISI) will be measured after two weeks of Dronabinol treatment.
  ISI ranges from 0 to 28, with higher scores indicating greater sleep disturbance.
Post-Traumatic Stress Disorder; PTSD checklist (PCL-5) | 2 weeks
  The change in Post-Traumatic Stress Disorder; PTSD checklist (PCL-5) will be measured after two weeks of Dronabinol treatment.
  PCL-5 scores range from 0 to 80, with higher scores indicating greater PTSD symptom severity.

CONTACTS AND LOCATIONS:
Overall Officials: Bharati Prasad, MD, Principal Investigator — Jesse Brown VA Medical Center, Chicago, IL
Locations (1):
- Jesse Brown VA Medical Center, Chicago, IL, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No